CLINICAL TRIAL: NCT03645148
Title: Safety, Tolerability and Partial Efficacy Study of a Personalized Neoantigen Cancer Vaccine in Treating Patients With Advanced Pancreatic Cancer
Brief Title: Clinical Study of a Personalized Neoantigen Cancer Vaccine in Treating Patients With Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Provincial People's Hospital (Other)
Collaborators: Hangzhou Neoantigen Therapeutics Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Liu Yang, MD, Zhejiang Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INEO-P-001
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Pancreatic Cancer; Pancreatic Carcinoma
Keywords: Neoantigen, Pancreatic Cancer, iNeo-Vac-P01,Peptide Vaccine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Colony-Stimulating Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iNeo-Vac-P01 (Experimental): Personal Cancer Vaccine: iNeo-Vac-P01 (peptides)+ GM-CSF;
  Peptides: 4 x 100 mcg per peptide given on days 1, 4, 8, 15, 22, 78, and 162 for a total of 7 doses;
  GM-CSF: 4 x 40 mcg (total dose 160 mcg) given on days 1, 4, 8, 15, 22, 78, and 162 for a total of 7 doses
  Interventions: Biological: iNeo-Vac-P01; Other: GM-CSF

INTERVENTIONS:
Biological: iNeo-Vac-P01 — Neoantigen peptides
Other: GM-CSF — immune adjuvant
  Other Names: granulocyte-macrophage colony stimulating factor

SUMMARY:
This research study is evaluating a new type of pancreatic cancer vaccine called "Personalized Neoantigen Cancer Vaccine" as a possible treatment for advanced pancreatic cancer. The purpose of the clinical study is evaluating the safety, tolerability and partial efficacy of the personalized neoantigen cancer vaccine in the treatment of Chinese patients with advanced pancreatic cancer, so as to provide a new personalized therapeutic strategy for advanced pancreatic cancer patients.

It is known that cancer patients have mutations (changes in genetic material) that are specific to an individual patient and tumor. These mutations can cause the tumor cells to produce proteins that appear very different from the body's own cells. It is possible that these proteins used in a vaccine may induce strong immune responses, which may help the participant's body fight any tumor cells that could cause the cancer to come back in the future. The study will examine the safety of the vaccine when given at several different time points and will examine the participant's blood cells for signs that the vaccine induced an immune response.

ELIGIBILITY:
Inclusion Criteria:

* Must freely sign informed consent;
* Aged 18 to 70 years old;
* The expected survival period is more than 6 months;
* ECOG score is 0 or 1;
* Advanced pancreatic cancer diagnosed by Pathology and imageology;
* Tumor cannot be excised by surgery, and multiline chemotherapy, radiation, targeted therapy fails, or other treatments cannot be tolerated;
* At least one measurable lesions;
* To be able to obtain sufficient tumor tissue samples and blood samples for analysis, or to have genomic/exon/transcriptional data of tumor tissues and normal tissues, and the data meet the analysis requirements;
* The main organs function is normal, such as the heart, liver and kidney;
* Haematological index:

neutrophil count≥1.5×10e9/L hemoglobin≥10g/dL platelet count≥100×10e9/L

* Biochemical index:

Total bilirubin is less than or equal to 1.5 times the upper limit of normal value (ULN) AST and ALT is less than or equal to 2.5 times the upper limit of normal value Serum creatinine and urea nitrogen (BUN) is less than or equal to 1.5 times the upper limit of normal value

* Pregnant, lactating women and women of child-bearing age must have a negative pregnancy test within 7 days before entering the group, and short-term have no fertility plan, and are willing to take protective measures (contraception or other birth control methods) before and during the clinical trial;
* Good compliance, able to follow research protocols and follow-up procedures.

Exclusion Criteria:

* Diagnosed as other malignant tumor;
* There have been bone marrow or stem cell transplants;
* No neoantigen was found in the sequencing data;
* Systemic cancer treatment or other drugs under study were treated within 4 weeks prior to Individualized tumor targeted polypeptides treatment;
* Received other polypeptide inoculation 4 weeks before treatment; Patients may not be vaccinated with other polypeptides 8 weeks after the last individualized tumor targeted polypeptides trentment;
* Active bacterial or fungal infections identified clinically (>= level 2 of NCI-CTC edition 3);
* Patients with HIV, HCV, HBV infection, severe asthma, autoimmune disease, immunodeficiency or treated with immunosuppressive drugs;
* Severe coronary or cerebrovascular disease, or other diseases that the investigators considered should to be exclusion;
* Drug abuse. Clinical, psychological or social factor result in affecting informed consent or research implementation;
* Have a history of drug or polypeptide allergies, or people who are allergic to other potential immunotherapies.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | 2 years
Number of participants experiencing clinical and laboratory adverse events (AEs) | 1 year

SECONDARY OUTCOMES:
Overall Survival Rate | 2 years
Progression Free Survival | 2 years

OTHER OUTCOMES:
Measurement of CD4/CD8 T lymphocyte subsets | 2 years
The polypeptide antigen - induced IFN-γ T cells responses | 2 years
Peripheral blood T cell receptor sequencing analysis | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Ott PA, Hu Z, Keskin DB, Shukla SA, Sun J, Bozym DJ, Zhang W, Luoma A, Giobbie-Hurder A, Peter L, Chen C, Olive O, Carter TA, Li S, Lieb DJ, Eisenhaure T, Gjini E, Stevens J, Lane WJ, Javeri I, Nellaiappan K, Salazar AM, Daley H, Seaman M, Buchbinder EI, Yoon CH, Harden M, Lennon N, Gabriel S, Rodig SJ, Barouch DH, Aster JC, Getz G, Wucherpfennig K, Neuberg D, Ritz J, Lander ES, Fritsch EF, Hacohen N, Wu CJ. An immunogenic personal neoantigen vaccine for patients with melanoma. Nature. 2017 Jul 13;547(7662):217-221. doi: 10.1038/nature22991. Epub 2017 Jul 5. PMID 28678778
- [Background] Weden S, Klemp M, Gladhaug IP, Moller M, Eriksen JA, Gaudernack G, Buanes T. Long-term follow-up of patients with resected pancreatic cancer following vaccination against mutant K-ras. Int J Cancer. 2011 Mar 1;128(5):1120-8. doi: 10.1002/ijc.25449. PMID 20473937
- [Derived] Chen Z, Zhang S, Han N, Jiang J, Xu Y, Ma D, Lu L, Guo X, Qiu M, Huang Q, Wang H, Mo F, Chen S, Yang L. A Neoantigen-Based Peptide Vaccine for Patients With Advanced Pancreatic Cancer Refractory to Standard Treatment. Front Immunol. 2021 Aug 13;12:691605. doi: 10.3389/fimmu.2021.691605. eCollection 2021. PMID 34484187